CLINICAL TRIAL: NCT06736119
Title: Effects of Task-oriented Intervention of Upper Limb on Coordination and In-hand Manipulation Among Children With Developmental Coordination Disorder
Brief Title: Effects of Task-Oriented Intervention in Children With Developmental Coordination Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0703
Record Dates: First submitted 2024-11-03; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Developmental Coordination Disorder
Keywords: Developmental Coordination Disorder; Task-Oriented Intervention; Upper limb
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: it will be qusai experimental study in which non-probability convenient sampling technique will be used. Interventional group of 4 to 12 age will be pormed in which participants will recieve task oriented interventions.
Masking Description: No one will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Task-oriented intervention (Experimental): task-oriented intervention for individual of developmental coordination disorder
  Interventions: Behavioral: Task Oriented Intervention

INTERVENTIONS:
Behavioral: Task Oriented Intervention — Intervention group will recieve task oriented interventions.Throwing and catching balls of different sizes and weights will be done. For writing, a task-oriented approach has 4 phases that will involve writing,correcting and fun writing 30-minute per session. Interventions provided 3 days per week for 3 months.

SUMMARY:
physical coordination is impacted by developmental coordination disorder (DCD), commonly referred to as dyspraxia. It makes a youngster appear to move clumsily and perform worse than expected in everyday tasks for their age. Fine and gross motor coordination issues are a hallmark of this neurodevelopmental disorder. Task-oriented therapies help children with DCD develop their skills, coordination, and manipulative abilities by including them in intentional, goal-directed tasks. This is noteworthy because a child's quality of life can be greatly impacted by these skills, which are essential for everyday tasks like writing, tying shoelaces, walking, and balance. The purpose of the research is to ascertain how task-oriented upper limb intervention affects children with impaired coordination and hand-eye coordination.

DETAILED DESCRIPTION:
The task-oriented intervention aimed at the upper limbs will be administered to the intervention group. For 3 months, interventions were offered 3 days a week.Over the course of 6 months, this quasi-experimental study will be carried out in Lahore. Data will be gathered from the Harbanspura branch of The Punjab School and the Askari School System in Mughalpura. There will be 18 students in the study. The study's inclusion criteria will be children with developmental coordination disorders between the ages of 4 and 12 Youngsters needed to be able to comprehend and adhere to instructions, both boys and girls who scored between 15 and 57 overall on the Developmental Coordination Disorder Questionnaire 2007.Children with congenital respiratory, cardiovascular, or musculoskeletal disorders, as well as those with unstable seizures, will be excluded. Both before and after the operation, data will be gathered. The Movement Assessment Battery for Children (MABC-2), the Developmental Coordination Disorder Questionnaire, and the ABIL HAND KID instrument will be used to assess subjects with developmental coordination disorders.

ELIGIBILITY:
Inclusion Criteria:

* Developmental coordination disorder children aged 4 to 12 years old.
* Have a total score of 15-57 on the Developmental Coordination Disorder Questionnaire2007.
* Children had to be able to understand and follow instructions.
* Boys and girls both are included

Exclusion Criteria:

* Children with unstable seizures will be excluded.
* DCD children with any congenital cardio-respiratory condition, congenital musculoskeletal condition.
* DCD children with severe visual and/or hearing disability preventing them from completing exercises prescribed by either program.
* Children with behavioral difficulty making them unable to complete exercises prescribed by either program

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-01-28 (Estimated); Study Completion 2025-02-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Motor Coordination as Measured by the DCDQ | 15 minutes
  The DCDQ evaluates changes in motor coordination in children aged 4-16 years based on parent-reported outcomes. It measures three subscales: Control During Movement, Fine Motor/Handwriting, and General Coordination. Scores are collected at pre and post-intervention (3 months), with higher scores indicating improved motor coordination.
Changes in Manual Ability Assessed by the ABILHAND-Kids Questionnaire | 10 minutes
  The ABILHAND-Kids Questionnaire evaluates changes in manual ability and bimanual coordination in daily activities among children with motor impairments. It is a parent-reported measure assessing the ease or difficulty with which a child performs 21 bimanual tasks in their daily life. Scores are collected at baseline (pre-intervention), and post-intervention (3 months), with higher scores indicating improved manual ability and functional performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mah Noor Fatima, MS*, Principal Investigator — Riphah International University
Locations (1):
- Askari School System, Mughalpura, The Punjab School Harbunspura baranch, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Civetta LR, Hillier SL. The developmental coordination disorder questionnaire and movement assessment battery for children as a diagnostic method in Australian children. Pediatr Phys Ther. 2008 Spring;20(1):39-46. doi: 10.1097/PEP.0b013e31815ccaeb. PMID 18300932